CLINICAL TRIAL: NCT03883893
Title: Randomized Prospective Study Investigating the Analgesic Efficacy of Intravenous Acetaminophen in Reducing Post-Tonsillectomy Pain in Pediatric Patients
Brief Title: IV Acetaminophen and Post-Tonsillectomy Pain
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Mentor for PI left institution. Study was not renewed.
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2018-0565
Record Dates: First submitted 2019-03-19; First posted 2019-03-21 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Tonsillectomy; Adenoidectomy
Keywords: Tonsillectomy; Intravenous Acetaminophen; Pediatric
MeSH Terms: interventions — Acetaminophen; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Clinical research coordinator, parent and participant will be masked until participant is discharged from hospital. OR staff will not be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IV Tylenol (Active Comparator): Participants will receive IV acetaminophen 15mg/kg in the OR.
  Interventions: Drug: Intravenous acetaminophen
- Normal Saline (Placebo Comparator): Participants will receive 0.9% normal saline in the OR. The amount received will be equivalent of what would be given if they were receiving IV acetaminophen.
  Interventions: Other: Normal saline

INTERVENTIONS:
Drug: Intravenous acetaminophen — Intravenous acetaminophen will be given in the OR.
  Other Names: IV Tylenol
  Arms: IV Tylenol
Other: Normal saline — Normal saline will given if randomized to this group.
  Arms: Normal Saline

SUMMARY:
This study is a randomized prospective study to compare the post-operative analgesic efficacy of intravenous acetaminophen 15 mg/kg to an equal volume of 0.9% normal saline when all other analgesic interventions have been standardized for all patients enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is age 3 to 10 years (inclusive)
2. The subject weighs more than 10.0 kg (inclusive of the tenth kilogram)
3. The subject is scheduled for the following: Elective tonsillectomy or tonsillectomy with adenoidectomy scheduled on an outpatient basis, with acceptable inclusion of patients also having PETs and/or EUA of ear
4. The subject is ASA patient classification I-II
5. The subject's legally authorized representative has given written informed consent to participate in the study and when appropriate, the subject has given assent or consent to participate.

Exclusion Criteria:

1. Additional surgical procedures are being performed concurrently;
2. The subject is ASA classification > II;
3. The subject has pre-existing allergy or known hypersensitivity to acetaminophen;
4. The subject receives midazolam as a premedication;
5. The subject has a history of chronic malnutrition;
6. The subject has any other condition, which in the opinion of the principal investigator, would not be suitable for participation in the study

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain scores | Every 5 minutes after awake in recovery room for 30 minutes
  FLACC (Face, Legs, Activity, Cry, Consolability) behavior scale Each area measured is graded 0 - 2 and then totaled. Total score will range from 0 - 10. A total score of 0 - patient is relaxed and comfortable, 1 - 3 - patient is mildly uncomfortable, 4 - 6 - patient is in moderate pain, 7 - 10 - patient is having severe discomfort/pain

SECONDARY OUTCOMES:
Quality of emergence from anesthesia | When first spontaneous eye movement occurs in recovery room
  Pediatric Anesthesia Emergence Delirium scale (PAED)
  This scale uses 5 criteria to determine the extent of emergence delirium in children. "The child makes eye contact with the caregiver", "The child's actions are purposeful", The child is aware of his/her surroundings", The child is restless" and "The child is inconsolable." Each of these 5 catagories are scored on a 0-4 scale. The higher the total number the greater the extent of the emergence delirium.

CONTACTS AND LOCATIONS:
Overall Officials: Judy Audas, APRN-CRNA,MSN, Principal Investigator — Children's Hospital Medical Center, Cincinnati